CLINICAL TRIAL: NCT00211666
Title: Improving the Delivery of Effective Care to Minorities
Brief Title: Improving Hypertension Control in East and Central Harlem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01HS010859-05 (AHRQ); 00-0053
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Hypertension; blood pressure; self management; nurse management; racial disparities; cardiovascular disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Nurse management, home blood pressure monitors, and a chronic disease self management course.

SUMMARY:
This hypertension project is evaluating strategies developed to target problems underlying lack of blood pressure control among treated but uncontrolled hypertensive patients in East and Central Harlem.

DETAILED DESCRIPTION:
The hypertension project will tailor improvement strategies to the problems identified as underlying underuse among treated but uncontrolled hypertensive patients in East and Central Harlem, New York City. Along with the communities' 6 major health providers, we will first combine qualitative and quantitative methods to identify specific patient, provider, and system problems, and customize interventions to address them. In a randomized controlled trial, we will then randomly assign 480 patients among 4 arms: nurse management, blood pressure monitors alone, usual care, and peer led chronic disease self-management course. During the 18-month trial, patients self-monitor their blood pressure or attend a self-management course, or nurse managers will assess patients' needs, counsel them, address any access barriers, and follow up with regular telephone contacts; convey information, including blood pressures from patients' self-monitoring, between patients and physicians to inform possible medication changes; and ameliorate any systems problems. We will assess differences in blood pressure reductions among the 4 arms as the primary outcome, and in quality of life, patient satisfaction, costs, and cost-effectiveness as secondary outcomes. The findings will provide new knowledge about the relationship between these changes and patient and clinician knowledge, attitudes, and behaviors. The educational course is designed to teach patients tools for managing their chronic illness which will empower them to improve their overall health and is specifically tailored for patients living with asymptomatic chronic illnesses and will emphasize communication with health care providers. In partnership with community organizations and the policymakers, we will disseminate successful findings within these communities and throughout the state and the nation.

ELIGIBILITY:
Inclusion Criteria:

Male and female, English or Spanish speaking African American and/or Hispanic patients with uncontrolled hypertension who have been seen in either the Cardiology clinic, Internal Medicine Associates (IMA) or Geriatric clinic at least twice in a given year at least 18 years of age.

Exclusion Criteria:

This study is about hypertension control among African Americans and Hispanics, these are the ethnic groups with disparities in CVD that we want to improve so other races are excluded. The study is for adults with hypertension; therefore, we are excluding anyone who is under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2002-09; Study Completion 2006-08

PRIMARY OUTCOMES:
Differences in blood pressure reduction among the four study arms.

SECONDARY OUTCOMES:
Quality of life
patient satisfaction
costs
cost-effectiness

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chassin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States